CLINICAL TRIAL: NCT06754020
Title: Application of Artificial Intelligence for Precision Medicine in TCM Tongue Diagnosis and Syndrome Differentiation in Myasthenia Gravis Compared to Healthy Controls
Brief Title: TCM Tongue Diagnosis and Syndrome Differentiation in Myasthenia Gravis Compared to Healthy Controls
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Ting Yeh (Other)
Responsible Party: Sponsor-Investigator, Yi Ting Yeh, Principal Investigator, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20221019R
Record Dates: First submitted 2024-08-08; First posted 2024-12-31 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; traditional Chinese medicine
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disease Group (Experimental): Participants with myasthenia gravis will be recruited and assessed in the Neurology Department's outpatient clinic and wards at Shin Kong Hospital.
  Interventions: Device: Heart Rate Variability,HRV - ANSWatch; Device: Traditional Chinese Medicine Tongue Imaging
- **Healthy Control Group** (Experimental): The healthy control group will be recruited from community settings and universities in Taipei City.
  Interventions: Device: Heart Rate Variability,HRV - ANSWatch; Device: Traditional Chinese Medicine Tongue Imaging

INTERVENTIONS:
Device: Heart Rate Variability,HRV - ANSWatch — Please have the participant lie down and rest for 10 minutes, and remove any metallic items from their body. Next, put on the wrist-worn monitor, and avoid moving during the monitoring process. The device will emit a sound when the monitoring session is complete.
Device: Traditional Chinese Medicine Tongue Imaging — Use a camera to capture images of the tongue, and then have a Traditional Chinese Medicine (TCM) practitioner perform the diagnosis based on these images.

SUMMARY:
Myasthenia gravis primarily results from neuromuscular junction dysfunction and damage, leading to chronic muscle weakness. While combined traditional and Western medicine treatments are now common, TCM tongue diagnosis remains a simple and practical clinical method. However, results can vary among different practitioners. Therefore, you are interested in using scientific methods to compare TCM tongue diagnosis images between patients with myasthenia gravis and healthy individuals to aid in diagnosis.

DETAILED DESCRIPTION:
In Taiwan, the prevalence of severe myasthenia gravis is approximately 14 per 100,000 people, with an incidence rate of about 2 per 100,000 people.

Currently, combined traditional and Western medicine treatments are very popular. In Traditional Chinese Medicine (TCM), tongue diagnosis is a simple and practical clinical method, focusing on aspects such as the tongue body, coating, color, and sublingual veins. Clinical evaluation often relies on the experience and knowledge of TCM practitioners, which can be influenced by subjective factors like diagnostic skills. As a result, findings may vary depending on the observer.

To improve diagnostic accuracy, using scientific methods to support TCM tongue diagnosis can provide more precise information for practitioners and enhance the clinical application value of tongue diagnosis in TCM.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with myasthenia gravis by a physician.
2. Able to understand and communicate in Mandarin and Taiwanese.
3. Cognitively alert and without a diagnosis of psychiatric disorders.
4. Willing to undergo tongue imaging and instrument measurements.

Exclusion Criteria:

1. Patients with severe organ diseases.
2. Hearing loss patients who are unable to complete the questionnaire.
3. Patients with aphasia who are unable to complete the questionnaire.
4. Have eaten food or drinks that can easily contaminate tongue coating within 2 hours.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-01-17 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
What are the differences in tongue diagnosis in traditional Chinese medicine between the disease group and the healthy population? | 2025/01/18 (4th week)
  Using a camera to capture images of the tongue, traditional Chinese medicine practitioners were invited to evaluate the tongue photographs. After organizing the data, a comparison between the two groups was conducted in the fourth week.

SECONDARY OUTCOMES:
Observe the differences in physical constitution and tongue diagnosis between patients with myasthenia and healthy people. | 2025/01/18 (4th week)
  The disease group and the control group were asked to complete the Traditional Chinese Medicine Constitution Questionnaire (TCMCQ) separately. After organizing the data, statistical analysis was conducted in the fourth week.

CONTACTS AND LOCATIONS:
Locations (1):
- Yi Ting Yeh, New Taipei City, Tamsui District, Taiwan